CLINICAL TRIAL: NCT05155982
Title: A Randomized, Observer-Blind, Dose-Escalation, Placebo-Controlled Phase 1 Clinical Trial of COVAC-1 in Generally Healthy Adults
Brief Title: A Clinical Trial of COVAC-1, a COVID-19 Vaccine, in Generally Healthy Adults
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Decided not to move forward with the study design.
Sponsor: University of Saskatchewan (Other)
Collaborators: Government of Canada (Other Government); Government of Saskatchewan (Other Government)
Responsible Party: Principal Investigator, Volker Gerdts, Director - Vaccine and Infectious Disease Organization, University of Saskatchewan
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: COVAC-002
Record Dates: First submitted 2021-11-30; First posted 2021-12-14 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2
MeSH Terms: interventions — COVAC-1 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Group A (18-54 yrs) (Experimental): COVAC-1 25 ug
  Interventions: Biological: COVAC-1
- Group B (18-54 yrs) (Placebo Comparator): Placebo Control
  Interventions: Biological: Saline Placebo
- Group C (18-54 yrs) (Experimental): COVAC-1 50 ug
  Interventions: Biological: COVAC-1
- Group D (18-54 yrs) (Placebo Comparator): Placebo Control
  Interventions: Biological: Saline Placebo
- Group E (55+ yrs) (Experimental): COVAC-1 25 ug
  Interventions: Biological: COVAC-1
- Group F (55+ yrs) (Placebo Comparator): Placebo Control
  Interventions: Biological: Saline Placebo
- Group G (55+ yrs) (Experimental): COVAC-1 50 ug
  Interventions: Biological: COVAC-1
- Group H (55+ yrs) (Placebo Comparator): Placebo Control
  Interventions: Biological: Saline Placebo

INTERVENTIONS:
Biological: COVAC-1 — Intramuscular vaccine against SARS-CoV-2
  Arms: Group A (18-54 yrs); Group C (18-54 yrs); Group E (55+ yrs); Group G (55+ yrs)
Biological: Saline Placebo — Intramuscular injection of saline placebo
  Arms: Group B (18-54 yrs); Group D (18-54 yrs); Group F (55+ yrs); Group H (55+ yrs)

SUMMARY:
VIDO has developed a vaccine called COVAC-1.

The study vaccine contains a portion of the SARS-CoV-2 spike protein, called S1. The spike protein is the part of the virus that is responsible for attaching to the surface of host cells. COVAC-1 contains an adjuvant called TriAdj. An adjuvant is a compound that is added to a vaccine to help the vaccine produce a better immune response. The TriAdj adjuvant is made up of three components (a toll-like receptor agonist polyI:C, an immunostimulatory host defense protein HDP IDR-1002 and a polyphosphazene carrier system, PCEP). The three components work together to improve the body's response to the S1 protein. The COVAC-1 vaccine is expected to stimulate the body to make antibodies against the S1 protein. The antibodies will recognize the viral spike protein if the body is exposed to the virus and prevent or reduce the severity of COVID-19 illness. In animal studies, the immune response generated by the COVAC-1 vaccine was able to protect the vaccinated animals against a severe SARS-CoV-2 infection.

Phase 1 is a multi-centred, multi-national trial of the COVAC-1 vaccine to be completed in Canada and Brazil. It will be a randomized, observer-blinded, and placebo-controlled study to assess the safety and immunogenicity of two dosing levels (25 and 50 µg S1 protein) administered twice (4 weeks apart) in healthy adults 18 through 54 years of age (Arm 1a) and 55 years of age and older (Arm 1b).

Enrolment and vaccination of participants will be staggered over time based on vaccine dose. Study participants aged 18 to 54 and those >55 years of age will commence in parallel at the starting dose of 25 ug and after approval by Sponsor based upon recommendations from the Data Safety Monitoring Board (DSMB), new study participants will be allowed to receive the higher dose of 50 ug. Approval will also be sought from Sponsor, based on recommendations provided by the DSMB, to proceed with the second dose in each dosing and age group.

Within the same age group, the 8 participants receiving the lower dose are randomized with 4 participants receiving placebo and the 8 participants receiving the highest dose are randomized with 4 participants receiving placebo.

Within each dose level of 12 participants, it is proposed to immunize a first cohort of 3 participants (including at least 2 active vaccine participants) and pending no holding rule is met after 48 hours, as determined by the 48-hour-post-dose 1 phone call, to immunize the remaining 9 participants within that dose level. Every attempt will be made to fully enroll all age groups.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy male and female adults aged 18 years of age or older at the time of signing the informed consent form (i.e., 18 to 54 for Arm 1a and ≥55 for Arm 1b);
2. Good general health as determined by screening evaluation no greater than 30 days before injection of first dose; Note: Participants who are overtly healthy as determined by medical evaluation or are considered medically stable according to the judgment of the Investigator. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months prior to enrolment, and/or hospitalization within the entire study period is not anticipated. Also, the participant appears likely to be able to remain in follow-up through the end of protocol-specified period. Mild to moderate well-controlled comorbidities are allowed.
3. If female of child-bearing potential and heterosexually active, practice of adequate contraception for 30 days prior to injection, negative pregnancy test on the day of injection, and agreement to continue adequate contraception until 180 days after the second injection and;
4. Written informed consent, after review of the consent form and having adequate opportunity to discuss the study with an Investigator or a qualified designee.

Exclusion Criteria:

1. Presence of any febrile illness or any known or suspected acute illness on the day of any immunization;
2. Any immunodeficiency (congenital or acquired) disease, disorder, or finding that may significantly increase the risk of study participant or, in the Investigator's judgment, make the participant inappropriate for the study;
3. Clinically significant bleeding disorder (e.g., clotting factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture;
4. Receiving systemic immunosuppressive therapy or history of receiving chemotherapy in last 5 years other than topical agents;
5. Receipt of systemic glucocorticoids (a dose ≥ 20 mg/day prednisone or equivalent for 14 days) within 1 month, or any other cytotoxic or immunosuppressive drug within 6 months prior to injection of first dose;
6. Cancer diagnosis in the last 5 years, excluding basal cell and squamous cell carcinoma of the skin, which are allowed;
7. Presence of autoimmune disease;
8. Receipt of any investigational drug within 6 months;
9. Receipt of any non-COVID-19 authorized vaccines within 2 weeks of receiving study dose injection;
10. Receipt of any authorized COVID-19 vaccine prior to study enrollment;
11. Receipt of any other experimental SARS-CoV-2/COVID-19 or other experimental coronavirus vaccine(s) at any time prior to or during the study;
12. Receipt of blood products or immunoglobulin (IVIg or IMIg) within 3 months of study entry/baseline serologic evaluation;
13. Current anti-tuberculosis therapy;
14. History of any reaction or hypersensitivity likely to be exacerbated by any component of the study vaccine;
15. Hematologic or biochemical laboratory abnormalities (blood or urine), as defined by lab normal ranges. To exclude transient abnormalities, the Investigator may repeat a test once, and if the repeat test is normal according to local reference ranges, participant may be enrolled. Grade 1 abnormalities of laboratory values will not be exclusionary if considered not clinically significant by the Investigator. And;
16. Known current or previous laboratory-confirmed SARS-CoV-1 OR SARS-CoV-2 infection, as documented by a positive polymerase chain reaction (PCR) test from a nasal swab OR known or laboratory-confirmed positive serology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events (AEs) from the first injection to Day 28, in all participants, in all groups | Day 0 - 28
  The occurrence of each solicited local and general AE, during each 7-day follow-up period after injection (e.g., the day of injection and 6 subsequent days).
  * The occurrence of any unsolicited AEs for the entire study period.
  * The occurrence of any hematological (hemoglobin level, WBC, lymphocyte, neutrophil, eosinophil, and platelet count) and biochemical (ALT, AST, BUN, and Cr) clinically significant laboratory abnormality through to Day 28 and;
  * The occurrence of any serious AEs (SAEs) medically attended events (MAE), or adverse event of special interest (AESI).
Occurrence of AEs from the second injection to Day 56 (28 days post injection), in all participants, in all groups | Day 28 - 56
  * The occurrence of solicited local and general AE, during each 7-day follow-up period after the second injection (e.g., the day of 2nd injection and 6 subsequent days);
  * The occurrence of any unsolicited AEs for the entire study period and;
  * The occurrence of any hematological (hemoglobin level, WBC, lymphocyte, neutrophil, eosinophil, and platelet count) and biochemical (ALT, AST, BUN, and Cr) clinically significant laboratory abnormality through to Day 42.

SECONDARY OUTCOMES:
Specific antibody response induced by the vaccine against the SARS-CoV-2 S protein as measured by ELISA or measured by Neutralization Assay | Days 14, 28, 35, 42, 56, 90, 120, and 365
  The immune response to the study vaccine, as measured by antibody (e.g., IgG and other isotypes) directed to Wuhan spike antigen or neutralizing antibodies
Specific cell-mediated immunity (CMI) response induced by the vaccine against the SARS-CoV-2 virus | Days 0, 14, 28, 35, 42, 120, and 365
  The immune response to the study vaccine, as measured by cell immune response markers in PBMCs

OTHER OUTCOMES:
The specific antibody response induced by the vaccine against the SARS-CoV-2 RBD protein as measured by ELISA | Days 0, 14, 28, 35, 42, 56, 90, 120, and 365
  The immune response to the study vaccine, as measured by antibody directed to RBD antigen
Specific neutralizing response induced by the vaccine against one or more Variant(s) of Concern | Days 0, 14, 28, 35, 42, 56, 90, 120, and 365
  • The immune response to the study vaccine, as measured by neutralizing antibodies against Variant(s) of Concern

CONTACTS AND LOCATIONS:
Overall Officials: Volker Gerdts, DVM, Study Director — University of Saskatchewan

IPD SHARING:
Plan to Share IPD: No